CLINICAL TRIAL: NCT05675462
Title: A Phase 1b Dose-escalation and Cohort-expansion Study of the Safety/Tolerability, and Efficacy of Oncolytic Virotherapy Plus PD-1 Inhibitor and Lenvatinib for Patients With Advanced Hepatocellular Carcinoma
Brief Title: Oncolytic Virotherapy Plus PD-1 Inhibitor and Lenvatinib as Second-line or Later Therapy in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTIONS-04
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H101 + Tislelizumab+ Lenvatinib (Experimental): (Dose escalation and cohort expansion) H101 administered by intratumoral injection in combination with Tislelizumab administered intravenously (IV), and Lenvatinib administered orally.
  H101 intratumorally injection starts at day 0. Tislelizumab plus lenvatinib will be initiated on day 1. Tislelizumab will be administered at 200 mg i.v. every 3 weeks plus a lenvatinib (bodyweight ≥ 60 kg, 12 mg; < 60 kg, 8 mg) orally daily every 3 weeks until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Oncorine; Drug: Tislelizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Oncorine — a modified human recombinant type 5 adenovirus with genetic modifications
  Other Names: H101
Drug: Tislelizumab — PD-1inhibitor
Drug: Lenvatinib — TKI

SUMMARY:
The objective of this study is to evaluate the safety/tolerability efficacy of oncolytic virotherapy combined with Tislelizumab plus lenvatinib as second-line or later therapy in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Recent studies have suggested that local destruction of tumor tissue by oncolytic virus induced activation and maturation of dendritic cells and tumor-specific T cells by cross-presentation of tumor antigens. While pd-1 blocking antibody interferes with PD-1 mediated T-cell regulatory signaling. And combination of pd-1 blocking antibody plus lenvatinib showed increased ORR in many types of human cancers. Therefore, the objective of this study is to evaluate the safety and efficacy of oncolytic virotherapy combined with Tislelizumab plus lenvatinib as second-line or later therapy in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Age ≥ 18 years at time of study entry.
3. Participants must have unresectable or metastatic histologically or cytologically confirmed hepatocellular carcinoma.
4. Participants must have failed 1 line of systemic regimens for advanced hepatocellular carcinoma due to disease progression or toxicity.
5. Patients had been refractory or intolerant to previous systemic chemotherapy (oxaliplatin-based chemotherapy), targeted therapy (eg, sorafenib or lenvatinib), or anti-PD-1 or anti-PD-L1 based regimen.
6. At least one measurable site of disease as defined by RECIST criteria with spiral CT scan or MRI.
7. Performance status (PS) ≤ 2 (ECOG scale).
8. Life expectancy of at least 12 weeks.
9. Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥75 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula )
10. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

1. History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
2. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
3. RFA and resection administered less then 4 weeks prior to study treatment start.
4. Radiotherapy administered less then 4 weeks prior to study treatment start.
5. Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
6. Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
7. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
8. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
9. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to:

   1. history of interstitial lung disease
   2. Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection)
   3. known acute or chronic pancreatitis
   4. active tuberculosis
   5. any other active infection (viral, fungal or bacterial) requiring systemic therapy
   6. history of allogeneic tissue/solid organ transplant
   7. diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Tislelizumab treatment.
   8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
   9. Live vaccine within 30 days prior to the first dose of Tislelizumab treatment or during study treatment.
   10. History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of Tislelizumab treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS
10. Medication that is known to interfere with any of the agents applied in the trial.
11. Any other efficacious cancer treatment except protocol specified treatment at study start.
12. Patient has received any other investigational product within 28 days of study entry.
13. Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.

Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 28 days
  The DLT assessment period is defined as: Day of Injection through 28 days post injection (Safety Follow Up). A DLT will be defined as any Grade 3 or higher adverse event, as assessed by the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Maximum tolerated dose | max 24 months
  A MTD is determined if any cohort experiences 2 subjects with DLT's. Safety
Adverse event (AE). | max 24 months
Treatment emergent adverse event(TEAE). | max 24 months
Serious adverse event (SAE). | max 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | max 24 months
  ORR according to RECIST 1.1
DoR | max 24 months
  Duration of Response
PFS | max 24 months
  Progression Free Survival
OS | max 42 months
  Overall survival
DCR | max 24 months
  disdisease control rate
Detection of systemic and local immune activation in tumors and peripheral blood mononuclear cell will be assessed by single cell RNA seq and/or bulk RNA seq. | max 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No